CLINICAL TRIAL: NCT05094635
Title: Characteristics of Immunogenicity Against SARS-CoV-2 in the Community With Home-quarantined Covid-19 Patients in Ho Chi Minh City, Vietnam
Brief Title: Immunogenicity Against SARS-CoV-2 in COVID-19 Close Contacts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Lan Ngoc Vuong, Head of Department of Obstetrics and Gynaecology; Dean, Faculty of Medicine, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 473/HDDD-DHYD
Record Dates: First submitted 2021-10-25; First posted 2021-10-26 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Vaccine Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum and DNA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 IgG II Quant — 3ml of blood samples are collected, contained in heparin-free tubes, and centrifuged. Blood serum samples are collected and stored at the -80 Celcius degree. SARS-CoV-2 IgG antibodies in human serum and plasma are detected using chemiluminescent microparticle immunoassay (CMIA) technology on the ARCHITECT I 1000r System. Quality Control procedures will take place once daily, with three levels: one negative control and two positive controls. Sample, SARS-CoV-2 antigen-coated paramagnetic microparticles, and assay diluent are combined and incubated. The SARS-CoV-2 IgG antibodies present in the sample bind to the antigen-coated microparticles. The resulting chemiluminescent reaction is measured as a relative light unit (RLU). There is a direct relationship between the titres of IgG antibodies to SARS-CoV-2 in the sample and the RLU detected by the system optics. Interpretation of Results: < 50.0 AU/mL, Negative, ≥ 50.0 AU/mL, Positive

SUMMARY:
This study will investigate the presence of SARS-CoV-2 neutralizing antibody and its association with demographic information, medical history of SARS-CoV-2 infected individuals, exposure history of close contacts, vaccination status, and compliance with the strategies for self-quarantine to prevent the transmission in the community where SARS-CoV-2 infected individuals were home-quarantined and treated.

DETAILED DESCRIPTION:
In the 4th outbreak of the covid-19 pandemic in Ho Chi Minh City since 27 April 2021, asymptomatic or mild covid-19 patients were self-quarantined and treated at home. This home care setting could yield risk of SARS-CoV-2 transmission from the index cases to the people living surroundings. Therefore, this study will be performed to investigate the immunogenicity against SARS-CoV-2 in household members or people lived in the same municipality with home-quarantined covid-19 patients.

All people over 18 years old, living in 2 blocks (V and Y) of Ngo Gia Tu apartment, which is located in District 10, Ho Chi Minh City, will be recruited into this study. A survey will be conducted using a questionnaire to collect the data related to the basic demographic information, medical history of SARS-CoV-2 infected individuals, exposure history of close contacts, vaccination status, and compliance with the strategies for self-quarantine to prevent the transmission in the community.

At the time of recruitment, Covid-19 rapid antigen detection tests using nasopharyngeal swabs will be performed for all study subjects. In addition, a total of 5mL of intravenous blood samples will be collected for serum extraction and DNA isolation. SARS-CoV-2 neutralizing antibody levels in serum samples will be evaluated by a surrogate virus neutralization test by using NeutraLISA kit® (Euroimmun, Luebeck, Germany). DNA will be isolated and stored for further use in investigating the association of ACE2 genetic polymorphisms with the prevalence of SARS-CoV-2 neutralizing antibodies.

ELIGIBILITY:
Inclusion Criteria:

* People who lived in the two blocks (V and Y) of Ngo Gia Tu apartment, located in District 10, Ho Chi Minh City, Vietnam, from July to September 2021
* 18 years of age and older
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* People who were diagnosed with primary or secondary immunodeficiencies induced by diseases or medical treatments (immunosuppressants, chemotherapy, radiation therapy, ect.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People 18 years of age and older, who lived in 2 blocks (V and Y) of Ngo Gia Tu apartment, located in District 10, Ho Chi Minh City, Vietnam, from July to September 2021
Sampling Method: Non-Probability Sample
Enrollment: 772 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 anti-RBD IgG concentration | Up to 1 week after examination
  SARS-CoV-2 anti-RBD IgG antibody concentration was reported after analysing the specimen

CONTACTS AND LOCATIONS:
Overall Officials: Tuan D Tran, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Medicine and Pharmacy, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No